CLINICAL TRIAL: NCT03636711
Title: Adherence to Anti-infectious Treatment Protocols in Emergencies and Short-term Hospitalization at the Infectious Disease Department"
Brief Title: Antibiotic Stewardship in Infectious Disease Departement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-24
Record Dates: First submitted 2018-07-09; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: • Patient admitted to emergency for infectious syndrome Description of antibiotic protocol, according to a syndromic approach will be performed
  Interventions: Other: antibiotic protocol, according to a syndromic approach

INTERVENTIONS:
Other: antibiotic protocol, according to a syndromic approach — Description of patients who benefited or not the antibiotic protocol, according to a syndromic approach and analysis of the causes of non-adherence to the protocols

SUMMARY:
Consensual antibiotic protocols have been developed and validated locally by infectious disease specialists, internists and emergency physicians, in order to encourage their compliance. A preliminary study was conducted from June 2015 to February 2016, including 622 patients admitted to the emergency department for infectious syndrome such as /

* Pneumoniae
* Urinary tract infection
* Cellulitis
* Meningitis
* Malaria
* Febrile neutropenia
* Febrile acute diarrhea
* Fever back to the tropics
* Angina
* sexually transmitted infection This prospective study will observe and analyze the adherence of prescribers to these protocols. With description of patients who benefited or not the antibiotic protocol, according to a syndromic approach and analysis of the causes of non-adherence to the protocols. In order to limit the length of stay and reduce the cost of hospitalization..

DETAILED DESCRIPTION:
Consensual antibiotic protocols have been developed and validated locally by infectious disease specialists, internists and emergency physicians, in order to encourage their compliance. A preliminary study was conducted from June 2015 (setting up protocols) to February 2016, including 622 patients admitted to the emergency department for infectious syndrome such as /

* Pneumoniae
* Urinary tract infection
* Cellulitis
* Meningitis
* Malaria
* Febrile neutropenia
* Febrile acute diarrhea
* Fever back to the tropics
* Angina
* sexually transmitted infection This prospective study will observe and analyze the adherence of prescribers to these protocols. With description of patients who benefited or not the antibiotic protocol, according to a syndromic approach and analysis of the causes of non-adherence to the protocols. In order to limit the length of stay and reduce the cost of hospitalization..

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to emergency for infectious syndrome
* Patient > 18 years old.
* Patient who accept to have his medical records reviewed for research.

Exclusion Criteria:

* Patient < 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present a infectious syndrom
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
List of Antibiotic treatment | up to 12 weeks
  Description of the prescribed antibiotic treatment depending of infectious syndrome: name, duration for each treatment during hospitalization
  Data will be collected in the medical files:
  * date of introduction of antibiotic treatment
  * withdrawal dates
  * stop dates
  * antibiotic classes
Adverse events | up to 12 weeks
  Description of the cause of non adherence to antibiotic treatment initiates at hospital admission of antibiotherapy:
  Data will be collected in the medical files of patients:
  events leading to withdrawal or stop treatment (insufficiency renal, allergic reaction ... etc) date of events aggravation or recovery

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France